CLINICAL TRIAL: NCT04701827
Title: Affective Disorders: Eliminate WArning Signs And REstore Functioning: AWARE
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20029748
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Mood Disorders; Activities of Daily Living; Quality of Life
Keywords: Bipolar disorder; Mental disorder
MeSH Terms: conditions — Mood Disorders; Bipolar Disorder; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): AWARE intervention
  Interventions: Combination Product: AWARE intervention
- Control group (No Intervention): Treatment as usual (consisting of the standard out-patient mental health service routines in The Capital Region of Denmark)

INTERVENTIONS:
Combination Product: AWARE intervention — Comprehensive 360 degrees intervention. The intervention targets multiple aspects of the described enhancers of functioning based on on the ICF Brief Core Set. 1) ADL ability as a part of carrying out daily routines 2) Mood symptoms, medication and side effects 3) Social, relatives and network 4) Physical health, including BMI, biomarkers and exercise5) Cognition, circadian rhythm measured as sleep quality, and coping (stress reduction).
  Arms: Intervention group

SUMMARY:
Affective disorders are associated with impaired functioning and quality of life, as well as comorbid somatic disorders and increased mortality. Despite different medical and psychological treatment options, the prognosis for affective disorder remains largely unchanged. Consequently, the field needs new intervention strategies especially targeting the patient groups having impaired functioning. The core idea of the AWARE project is to focus on improving functioning and quality of life in patients with affective disorders every-day life using a comprehensive 360 degrees intervention.

The trial has a randomized, controlled, parallel-group design. Study participants will be 140 outpatients, male or female age 18-65 with a diagnosis of bipolar disorder or unipolar disorder, in a current state of remission, with an objectively rated impaired functioning. Participant will be randomized to six month AWARE intervention or treatment as usual (TAU).

Assessments encompassing Activities of Daily Living (ADL), neuropsychological testing, mood ratings, physical health and questionnaires on subjective cognitive complaints, psychosocial functioning, quality of life are, sleep quality and satisfaction with psychiatric treatment are carried out at baseline and after the end of treatment.

Discussion: It is hypothesised that the AWARE arm in comparison with standard care will improve observed ability to perform Activities of Daily Living (ADL) and improve Quality of Life.

DETAILED DESCRIPTION:
Despite different medical and psychological treatment options, the prognosis for affective disorder remains largely unchanged. Consequently, the field needs new intervention strategies especially targeting the patient groups having impaired functioning.

The core idea in the AWARE project is to focus on improving functioning and quality of life in patients with affective disorders every-day life using a comprehensive 360 degrees intervention. The present AWARE intervention represent an integrated treatment avenue to improve functioning in patients with affective disorders.

The aim of the study is, in a pragmatically Randomised Controlled Trial (RCT), to investigate the effect of a 360 degrees intervention based on the ICF Brief Core Set for BD and unipolar disorder targeting functioning.

The participants will upon inclusion, be randomised to participate in either 6 months AWARE treatment or standard care. The control group will receive standard care consisting of the standard out-patient mental health service routines in The Capital Region of Denmark.

The AWARE intervention targets multiple aspects of the described enhancers of functioning based on on the ICF Brief Core Set, including ADL ability as a part of carrying out daily routines.

The study carried out in a randomized design. The investigators who assess the patients are blinded to whether the patient has participated in the active or passive treatment arm, so the results will be valid. In addition, validated standardized survey methods according to all the outcomes is applied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder or unipolar disorder by ICD-10 diagnostic criteria (confirmed with a diagnostic interview), in a current state of remission (defined as HDRS-17 and YMRS scores of ≤ 14)
* At inclusion participants must have objectively rated impaired functioning defined as a score ≥ 11 according to the Functioning Assessment Short Test (FAST).
* Participants must be able to participate in 2/3 of the planned visits.

Exclusion Criteria:

* Severe somatic disorder interfering with daily living
* Ongoing alcohol or substance abuse
* Dementia or inability to cooperate with the study, including inability to speak and read Danish.
* ECT treatment within last 3 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
ADL ability | 6 month
  Assessment of Motor and Process Skills (AMPS) is a standardized observation-based assessment providing measures of the quality of ADL task performance.

SECONDARY OUTCOMES:
Patient quality of Life | 6 month
  PSS (Cohen's Perceived Stress Scale) and WHOQoL (World Health Organization, Quality of life)
Daily functioning | 6 month
  FAST (Functioning Assessment Short Test) and WHODAS (WHO Disability Assessment Schedule 2.0)

OTHER OUTCOMES:
Cognitive scores using a composite score from baseline to endpoint and physical health | 6 month
  SCIP, DART and Trailmaiking

CONTACTS AND LOCATIONS:
Overall Officials: Maj Vinberg, Prof, MD, DMSc, Study Director — Psychiatric Centre North Zealand, Copenhagen University Hospital
Locations (1):
- Psychiatric Centre North Zealand, Copenhagen University Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.
Time Frame: No current time frame
Access Criteria: Reasonable request

REFERENCES:
- [Derived] Schwarz R, Miskowiak KW, Christensen MS, Kessing LV, Vinberg M. Affective disorders: eliminate WArning signs And REstore functioning: AWARE. Results from a randomized controlled multimodular intervention study targeting functioning in patients with affective disorders. Psychol Med. 2024 Oct 31;54(14):1-10. doi: 10.1017/S0033291724002526. Online ahead of print. PMID 39479758
- [Derived] Schwarz R, Decker L, Seeberg I, Miskowiak KW, Kessing LV, Vinberg M. Affective disorders: eliminate WArning signs and REstore functioning-AWARE-a randomised controlled multimodule intervention study, presentation of design and intervention. BMJ Open. 2022 May 26;12(5):e058839. doi: 10.1136/bmjopen-2021-058839. PMID 35618335